CLINICAL TRIAL: NCT01321463
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of Once-Daily Orally Administered PH-797804 For 12 Weeks In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease (COPD) On A Background Of Salmeterol Xinafoate/ Fluticasone Propionate Combination
Brief Title: Study To Evaluate The Efficacy And Safety Of PH-797804 For 12 Weeks In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease (COPD) Taking Salmeterol Xinafoate/Fluticasone Propionate Combination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6631029
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — PH 797804

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PH-797804 (Experimental)
  Interventions: Drug: PH-797804
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PH-797804 — 6 mg oral tablet once daily for 12 weeks
  Arms: PH-797804
Drug: Placebo — Placebo oral tablet once daily for 12 weeks
  Arms: Placebo

SUMMARY:
PH-797804 is an oral ant-inflammatory drug that may reduce the inflammation that is associated with COPD. PH-797804 will be dosed to patients with COPD to evaluate its potential safety and efficacy profile in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including, the ages of 40 and 80 years.
* Subjects with a diagnosis, for at least 6 months, of moderate to severe COPD (GOLD) and who meet the criteria for Stage II-III disease.
* Subjects must have a smoking history of at least 10 pack-years and be current smokers or ex-smokers that gave up > 6 months ago.
* Subjects must be treated with a LABA/ICS combination for at least 1 month prior to screening.

Exclusion Criteria:

* A COPD exacerbation requiring treatment with oral steroids or hospitalization for the treatment of COPD within 3 months of screening.
* History or presence of significant cardiovascular disease.
* ECG abnormalities.
* Significant concomitant clinical disease that could interfere with the conduct, safety or interpretation of results of this study.
* Evidence of organ or blood disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Spirometry measures during 12 weeks of treatment and up to 2 weeks post treatment. | 12 Weeks

SECONDARY OUTCOMES:
Safety and tolerability measures (AEs, 12-lead ECG, lab safety) during 12 weeks of treatment and up to 2 weeks post treatment. | 12 Weeks
Dyspnea index scores. | 12 Weeks
Rescue bronchodilator usage. | 12 Weeks
Symptom scores. | 12 Weeks
Global impression of change (patient and clinician). | 12 Weeks
Blood sample for pharmacokinetics. | 12 Weeks
Blood and urine sample for biomarkers and molecular profiling. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (70):
- United States (20):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Trinity, Florida
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Duluth, Georgia
  - Pfizer Investigational Site, Norcross, Georgia
  - Pfizer Investigational Site, Livonia, Michigan
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, McKinney, Texas
- Argentina (3):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
- Australia (2):
  - Pfizer Investigational Site, Daw Park, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia
- Bulgaria (4):
  - Pfizer Investigational Site, Rousse
  - Pfizer Investigational Site, Sevlievo
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
- Canada (6):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Niagara Falls, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
- Chile (2):
  - Pfizer Investigational Site, Quillota, Región de Valparaíso
  - Pfizer Investigational Site, Valparaíso, Región de Valparaíso
- Czechia (5):
  - Pfizer Investigational Site, Kutná Hora
  - Pfizer Investigational Site, Liberec
  - Pfizer Investigational Site, Pardubice
  - Pfizer Investigational Site, Praha 10- Malesice
  - Pfizer Investigational Site, Tábor
- Hungary (4):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Szeged
  - Pfizer Investigational Site, Szombathely
- India (3):
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
- New Zealand (2):
  - Pfizer Investigational Site, Newtown
  - Pfizer Investigational Site, Tauranga
- Poland (3):
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zawadzkie
  - Pfizer Investigational Site, Łęczna
- Slovakia (6):
  - Pfizer Investigational Site, Bojnice
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Liptovský Hrádok
  - Pfizer Investigational Site, Považská Bystrica
  - Pfizer Investigational Site, Spišská Nová Ves
- South Africa (5):
  - Pfizer Investigational Site, Bellville, Cape Town
  - Pfizer Investigational Site, Tygerberg Campus, Cape Town
  - Pfizer Investigational Site, eManzimtoti, Durban
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Bloemfontein
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Stockholm
- United Kingdom (2):
  - Pfizer Investigational Site, Cottingham, Hull
  - Pfizer Investigational Site, Glasgow

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631029&StudyName=Study%20To%20Evaluate%20The%20Efficacy%20And%20Safety%20Of%20PH-797804%20For%2012%20Weeks%20In%20Adults%20With%20Moderate%20To%20Severe%20Chronic%20Obstructive%20Pulmonary%20